CLINICAL TRIAL: NCT00027846
Title: A Phase II Trial of Conformal Radiation Therapy for Pediatric Patients With Localized Ependymoma, Chemotherapy Prior to Second Surgery for Incompletely Resected Ependymoma and Observation for Completely Resected, Differentiated, Supratentorial Ependymoma
Brief Title: Observation or Radiation Therapy and/or Chemotherapy and Second Surgery in Treating Children Who Have Undergone Surgery for Ependymoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0121; CDR0000069086 (Other: Clinical Trials.gov); NCI-2012-02431 (Other: NCI); COG-ACNS0121 (Other: Children's Oncology Group)
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2017-01

CONDITIONS: Brain Tumor; Central Nervous System Tumor
Keywords: childhood supratentorial ependymoma; newly diagnosed childhood ependymoma; childhood infratentorial ependymoma
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cyclophosphamide; Etoposide; Podophyllotoxin; Vincristine; Radiotherapy; Radiation; Therapeutics; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GTR1 Differentiated Histology Supratentorial (Group 1) (No Intervention): Patients undergo observation.
- Radiation (Group 2) (Experimental): Supratentorial Anaplastic Ependymoma (GTR1, GTR2, NTR) and Anaplastic or Differentiated Infratentorial Ependymoma (GTR1, GTR2, NTR) and Supratentorial Differentiated Ependymoma(GTR2, NTR). Patients undergo conformal radiation therapy to the brain once daily 5 days a week for 6-6½ weeks.
  Interventions: Radiation: radiation therapy
- Sub-Total Resection Any Histology or Location (STR) (Group 3) (Experimental): Patients receive an initial course of chemotherapy comprising vincristine sulfate IV on days 1 and 8, carboplatin IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on days 1 and 2. Patients also receive filgrastim (G-CSF) subcutaneously or IV beginning on day 3 and continuing until blood counts recover. Patients then receive a second course of chemotherapy comprising vincristine sulfate IV on days 1 and 8, carboplatin IV over 1 hour on day 1, and oral etoposide on days 1-21. After completion of chemotherapy, patients are evaluated for second therapeutic conventional surgery. Patients who have unresectable disease undergo conformal radiation therapy. Patients who have resectable disease undergo second surgery followed by conformal radiotherapy.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cyclophosphamide; Drug: etoposide; Drug: vincristine sulfate; Radiation: radiation therapy; Drug: Mesna; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Biological: filgrastim — Given IV or SC (5mcg/kg/day) start on Day 3 and continue until ANC >1500/μl given subcutaneously or intravenously.
  Other Names: G CSF, G-CSF, granulocyte colony stimulating factor, granulocyte colony-stimulating factor
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)
Drug: carboplatin — Given IV (375 mg/m2/day) Day 1 given as an IV infusion over one hour. For patients with BSA <0.45m2 the dose is 12.5 mg/kg/day.
  Other Names: Blastocarb, Carboplat, Carboplatin Hexal, Carboplatino, Carbosin, Carbosol, Carbotec, CBDCA,
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)
Drug: cyclophosphamide — Given IV (1000mg/m2/day) Day 1 and 2 given as an IV infusion over one hour following carboplatin administration. For patients with BSA<0.45m2 the dose is 33mg/kg/day on Day 1 and 2.
  Other Names: Neosar, Procytox, Sendoxan, Syklofosfamid, WR-138719, Zytoxan
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)
Drug: etoposide — Given orally (50 mg/m2/day) orally once daily on Days 1 through 21. For patients with BSA < 0.45 m2, the dosage is 1.7 mg/kg/day on Days 1 through 21.
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside, EPEG, epipodophyllotoxin, Lastet, Toposar, VePesid
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)
Drug: vincristine sulfate — Given IV or orally (1.5mg/m2/day) (maximum dose 2 mg) Day 1 and 8 given as IV bolus. For patients with BSA<0.45m2 the dose is 0.05mg/kg.
  Other Names: 22-oxovincaleukoblastine, 57-22-7, leurocristine sulfate, VCR, Vincasar PFS
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)
Radiation: radiation therapy — Given once daily 5 days a week for 6-6½ weeks
  Other Names: irradiation, radiotherapy, therapy, radiation
  Arms: Radiation (Group 2); Sub-Total Resection Any Histology or Location (STR) (Group 3)
Drug: Mesna — Mesna (200mg/m2/dose) Day 1 and 2. For patients with BSA<0.45m2 the dose is (7mg/kg/dose). Combine mesna (200mg/m2) with cyclophosphamide and administer intravenously over one hour followed by mesna (200mg/m2) in 375 cc/m2 D5-1/2NS and run intravenously over 3 hours at 125cc/m2/hr. After 3 hour mesna, administer mesna (200 mg/m2/dose) IV over 15 minutes at hour 5.
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)
Procedure: therapeutic conventional surgery
  Arms: Sub-Total Resection Any Histology or Location (STR) (Group 3)

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to determine the effectiveness of specialized radiation therapy either alone or after chemotherapy and second surgery in treating children who have undergone surgery for localized ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the local control and pattern of failure in children with completely resected, differentiated, supratentorial localized ependymoma after initial surgical resection alone.
* Determine the rate of complete resection with second surgery after chemotherapy in patients with initially incompletely resected localized ependymoma.
* Determine the local control and pattern of failure in patients treated with conformal radiotherapy.
* Determine the influence of histologic grade on the time to progression in patients after treatment with conformal radiotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to extent of prior surgical resection.

* Group 1 (patients with supratentorial differentiated ependymoma who have undergone gross total resection and have no visible residual tumor): Patients undergo observation.
* Group 2 (patients with supratentorial anaplastic ependymoma or infratentorial anaplastic or differentiated ependymoma who have undergone gross total resection or near total resection): Patients undergo conformal radiotherapy to the brain once daily 5 days a week for 6-6½ weeks.
* Group 3 (patients with tumor of any histology or location who have undergone subtotal resection): Patients receive an initial course of chemotherapy comprising vincristine IV on days 1 and 8, carboplatin IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on days 1 and 2. Patients also receive filgrastim (G-CSF) subcutaneously or IV beginning on day 3 and continuing until blood counts recover. Patients then receive a second course of chemotherapy comprising vincristine IV on days 1 and 8, carboplatin IV over 1 hour on day 1, and oral etoposide on days 1-21. After completion of chemotherapy, patients are evaluated for second surgery. Patients who have unresectable disease undergo conformal radiotherapy. Patients who have resectable disease undergo second surgery followed by conformal radiotherapy.

Patients are followed every 4 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 250-350 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intracranial ependymoma

  * Differentiated ependymoma or anaplastic ependymoma
* No primary spinal cord ependymoma, myxopapillary ependymoma, subependymoma, ependymoblastoma, or mixed glioma
* No evidence of noncontiguous spread beyond primary site
* Initial surgical resection within the past 56 days

PATIENT CHARACTERISTICS:

Age:

* 1 to 21

Performance status:

* No restrictions

Life expectancy:

* At least 2 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Able to undergo MRI
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior or concurrent corticosteroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* More than 1 prior surgery allowed

Other:

* No other prior treatment for ependymoma

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 378 (Actual)
Dates: Start 2003-08; Primary Completion 2010-01-01 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Merchant, DO, PhD, Study Chair — St. Jude Children's Research Hospital
Locations (165):
- United States (140):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Maine Children's Cancer Program at Barbara Bush Children's Hospital, Scarborough, Maine
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Hospital, Newcastle, New South Wales
  - Prince of Wales Private Hospital, Randwick, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Herston, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- University Medical Center Groningen, Groningen, Netherlands
- Starship Children's Health, Auckland, New Zealand
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

RESULTS

PARTICIPANT FLOW:
Groups:
- Sub-Total Resection Any Histology or Location (STR) (Group 3): Patients receive initial course of chemotherapy comprising vincristine sulfate IV on days 1 and 8, carboplatin IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on days 1 and 2. Patients also receive filgrastim (G-CSF) subcutaneously or IV beginning on day 3 and continuing until blood counts recover. Patients then receive a second course of chemotherapy comprising vincristine sulfate IV on days 1 and 8, carboplatin IV over 1 hour on day 1, and oral etoposide on days 1-21. After completion of chemotherapy, patients are evaluated for second therapeutic conventional surgery. Patients who have unresectable disease undergo conformal radiation therapy. Patients who have resectable disease undergo second surgery followed by conformal radiotherapy.
  filgrastim: Given IV or SC (5mcg/kg/day) start on Day 3 and continue until ANC >1500/μl given subcutaneously or intravenously.
  carboplatin: Given IV (375 mg/m2/day) Day 1 given as an IV infusion over one hour. For patient
Period: Overall Study
Arm/Group | GTR1 Differentiated Histology Supratentorial (Group 1) | Radiation (Group 2) | Sub-Total Resection Any Histology or Location (STR) (Group 3)
Started | 13 | 287 | 78
Completed | 11 | 219 | 41
Not Completed | 2 | 68 | 37
Not completed — Lost to Follow-up | 0 | 41 | 9
Not completed — Withdrawal by Subject | 0 | 14 | 7
Not completed — Ineligible for study | 2 | 6 | 14
Not completed — Entry into another COG therapeutic study | 0 | 5 | 2
Not completed — Neuraxis dissemination during/after ther | 0 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GTR1 Differentiated Histology Supratentorial (Group 1) | Radiation (Group 2) | Sub-Total Resection Any Histology or Location (STR) (Group 3) | Total
Number analyzed (Participants) | 13 | 287 | 78 | 378
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 281 | 76 | 370
  Between 18 and 65 years | 0 | 6 | 2 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 10.78 [1.49 to 16.71] | 5.58 [1.01 to 21.01] | 5.18 [1.01 to 19.60] | 5.60 [1.01 to 21.01]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 114 | 38 | 159
  Male | 6 | 173 | 40 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 36 | 16 | 52
  Not Hispanic or Latino | 10 | 242 | 59 | 311
  Unknown or Not Reported | 3 | 9 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 15 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 1 | 34 | 4 | 39
  White | 9 | 219 | 62 | 290
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 3 | 14 | 5 | 22
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 28 | 8 | 37
  Netherlands | 0 | 6 | 3 | 9
  United States | 12 | 243 | 62 | 317
  Australia | 0 | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Event-free survival is calculated from the date of study enrollment to the date of disease progression, disease relapse, occurrence of second neoplasm, or death from any cause. The product-limit (Kaplan-Meier) estimate is for estimation of Event -free survival (EFS) probability at 5 years.
Time Frame: Up to 5 years after completion of study treatment
Population: The product-limit (Kaplan-Meier) estimate is for estimation of event-free survival probability at 5 years. All eligible patients in the study were included.
Measure: Number (95% Confidence Interval); unit: Probability of EFS at 5 years
Arm/Group | GTR1 Differentiated Histology Supratentorial (Group 1) | Radiation (Group 2) | Sub-Total Resection Any Histology or Location (STR) (Group 3)
Number analyzed (Participants) | 11 | 281 | 64
Probability of EFS at 5 years | 0.614 [0.33 to 0.90] | 0.685 [0.63 to 0.74] | 0.372 [0.25 to 0.50]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is measured from the date of study enrollment to the date to death. The product-limit (Kaplan-Meier) estimate is for estimation of OS probability at 5 years.
Time Frame: Up to 5 years after completion of study treatment
Population: All eligible patients in the study were included. The product-limit (Kaplan-Meier) estimate is for estimation of OS probability.
Measure: Number (95% Confidence Interval); unit: Probability of OS at 5 years
Arm/Group | GTR1 Differentiated Histology Supratentorial (Group 1) | Radiation (Group 2) | Sub-Total Resection Any Histology or Location (STR) (Group 3)
Number analyzed (Participants) | 11 | 281 | 64
Probability of OS at 5 years | 1 [1 to 1] | 0.862 [0.82 to 0.91] | 0.702 [0.58 to 0.82]

3. Secondary Outcome: Rate of Gross-total or Near-total Resection and Second Surgery After Chemotherapy
Description: The Rate Of Gross-Total or Near-Total Resection With Second Surgery After Chemotherapy Treatment.
Time Frame: At the time of second surgery
Population: Of 64 eligible patients in this group, 25 patients after chemotherapy had the second surgery. Of 25 patients with second surgery after chemotherapy, 19 had a Gross-Total or Near-Total resection. 19/25=76%.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sub-Total Resection Any Histology or Location (STR) (Group 3)
Number analyzed (Participants) | 25
percentage of participants | 76 [54.9 to 90.6]

4. Secondary Outcome: Event-free Survival (EFS)
Description: EFS between centrally reviewed differentiated ependymoma and anaplastic ependymoma for the patients who had sub-total resection initially. The event-free survival (EFS) defined as the date of disease progression, disease relapse, occurrence of a second neoplasm, or death from any cause, measured from the start date of radiation therapy. The product-limit (Kaplan-Meier) estimate is for estimation of EFS probability.
Time Frame: At 5 years since the time of radiation therapy.
Population: Of 64 eligible patients who had initial subtotal resection, 5 patients were off-therapy prior to radiation therapy, and 4 patients had a disease progression prior to radiation therapy. There were 55 eligible patients included in the analysis. The product-limit (Kaplan-Meier) estimate is for estimation of EFS probability.
Measure: Number (95% Confidence Interval); unit: Probability of EFS at 5 years
Groups:
- Differentiated Ependymoma: Differentiated ependymoma:tumor pathology by central review.
- Anaplastic Ependymoma: Anaplastic ependymoma:tumor pathology by central review.
Arm/Group | Differentiated Ependymoma | Anaplastic Ependymoma
Number analyzed (Participants) | 41 | 14
Probability of EFS at 5 years | 0.424 [0.27 to 0.58] | 0.298 [0.05 to 0.54]

5. Secondary Outcome: Event-free Survival (EFS)
Description: EFS between centrally reviewed differentiated ependymoma and anaplastic ependymoma for the patients who were treated with radiation therapy only. The event-free survival (EFS) defined as the time to disease progression, disease relapse, occurrence of a second neoplasm, or death from any cause, measured from the start of radiation therapy. The product-limit (Kaplan-Meier) estimate is for estimation of EFS probability at 5 years.
Time Frame: At 5 years since the time of radiation therapy
Population: Supratentorial Anaplastic Ependymoma (GTR1, GTR2, NTR) and Anaplastic or Differentiated Infratentorial Ependymoma (GTR1, GTR2, NTR) and Supratentorial Differentiated Ependymoma(GTR2, NTR). Patients undergo conformal radiation therapy to the brain once daily 5 days a week for 6-6½ weeks.
Measure: Number (95% Confidence Interval); unit: Probability of EFS at 5 years
Arm/Group | Differentiated Ependymoma | Anaplastic Ependymoma
Number analyzed (Participants) | 157 | 124
Probability of EFS at 5 years | 0.746 [0.68 to 0.82] | 0.607 [0.51 to 0.70]

6. Secondary Outcome: Local Control and Patterns of Failure
Description: Documented and analyzed qualitatively and quantitatively.
Time Frame: Up to 5 years after completion of study treatment
Population: All eligible patients in the study were included.
Measure: Number; unit: Participant
Arm/Group | GTR1 Differentiated Histology Supratentorial (Group 1) | Radiation (Group 2) | Sub-Total Resection Any Histology or Location (STR) (Group 3)
Number analyzed (Participants) | 11 | 281 | 64
Participant
  Local control | 6 | 217 | 29
  Pattern of failure local | 4 | 57 | 31
  Pattern of failure Metastatic | 0 | 26 | 5
  Pattern of failure local & metastatic | 1 | 7 | 4

ADVERSE EVENTS:
Description: All eligible patients were considered in the evaluation of adverse events. 281 eligible patients were in the group 2 and 64 eligible patients were in the group 3.
  GTR1 Differentiated Histology Supratentorial (Group 1) is an observation arm. Adverse events were not collected for the " GTR1 Differential Histology Supratentorial(Group 1)" observation arm..
Arm/Group | Radiation (Group 2) | Sub-Total Resection Any Histology or Location (STR) (Group 3)
Serious Adverse Events (participants affected / at risk) | 38/281 | 55/64
Other Adverse Events (participants affected / at risk) | 52/281 | 27/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation (Group 2) (N=281) | Sub-Total Resection Any Histology or Location (STR) (Group 3) (N=64)
Inner ear/hearing (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 0 (0) | 28 (31)
Hemolysis (e.g., immune hemolytic anemia, drug related hemolysis, other) (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Leukocytes (total WBC) (Investigations) | 4 (4) | 40 (47)
Lymphopenia (Investigations) | 8 (8) | 15 (18)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 (6) | 40 (49)
Platelets (Investigations) | 0 (0) | 25 (28)
Transfusion: Platelets (Blood and lymphatic system disorders) | 0 (0) | 10 (11)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1) | 14 (17)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 0 (0) | 1 (2)
Cardiovascular/General - Other (Specify) (Cardiac disorders) | 1 (1) | 0 (0)
Partial thromboplastin time (PTT) (Investigations) | 0 (0) | 2 (2)
Constitutional Symptoms - Other (Specify) (General disorders) | 1 (1) | 1 (1)
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound-infectious (Infections and infestations) | 1 (1) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (inflammation of cecum) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastrointestinal - Other (Specify) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1 (2) | 0 (0)
Alkaline phosphatase (Investigations) | 1 (1) | 0 (0)
SGOT (AST) (Investigations) | 1 (1) | 0 (0)
SGPT (ALT) (Investigations) | 1 (1) | 1 (2)
Catheter-related infection (Infections and infestations) | 1 (1) | 3 (5)
Febrile neutropenia (fever unknown origin no clinically or microbiologically documented infection) (Blood and lymphatic system disorders) | 1 (1) | 12 (13)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 2 (2) | 10 (10)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 3 (4)
Infection without neutropenia (Infections and infestations) | 9 (9) | 10 (13)
Amylase (Investigations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lipase (Investigations) | 0 (0) | 1 (9)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (<3yrs of age) (General disorders) | 0 (0) | 1 (1)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Mood alteration-depression (Psychiatric disorders) | 1 (1) | 0 (0)
Neuropathy - cranial (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy - motor (Nervous system disorders) | 1 (1) | 0 (0)
Personality/behavioral (Psychiatric disorders) | 2 (2) | 0 (0)
Seizure(s) (Nervous system disorders) | 3 (3) | 2 (2)
Neurology - Other (Specify) (Nervous system disorders) | 0 (0) | 1 (1)
Ocular/Visual - Other (Specify) (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation (Group 2) (N=281) | Sub-Total Resection Any Histology or Location (STR) (Group 3) (N=64)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Leukocytes (total WBC) (Investigations) | 16 (18) | 8 (9)
Platelets (Investigations) | 0 (0) | 7 (7)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 0 (0) | 6 (9)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 109/L) (General disorders) | 0 (0) | 5 (6)
Weight loss (Investigations) | 0 (0) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6)
Vomiting (Gastrointestinal disorders) | 19 (19) | 7 (9)
SGOT (AST) (Investigations) | 0 (0) | 6 (6)
SGPT (ALT) (Investigations) | 0 (0) | 7 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain sponsor approval.